CLINICAL TRIAL: NCT00613054
Title: Phase I Study of Zactima (ZD6474) Plus Imatinib Mesylate and Hydroxyurea for Patients With Recurrent Malignant Glioma
Brief Title: Ph I Zactima + Imatinib Mesylate & Hydroxyurea for Pts w Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Annick Desjardins (Other)
Collaborators: Novartis Pharmaceuticals (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Annick Desjardins, Assistant Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000393
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: GBM; Brain tumor; Zactima; Gleevec; Hydroxyurea; Glioblastoma; Gliosarcoma; Recurrent malignant glioma; ZD6474; Malignant glioma; Imatinib; Droxia; Hydrea; Hydroxycarbamide; Vandetanib
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms; Glioma | interventions — vandetanib; Imatinib Mesylate; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zactima + Gleevec + Hydrea (Experimental)
  Interventions: Drug: Zactima, Gleevec, Hydroxyurea

INTERVENTIONS:
Drug: Zactima, Gleevec, Hydroxyurea — Pts will start treatment on day 1 of cycle 1 w Zactima, imatinib mesylate & hydroxyurea. All 3 agents administered in continuous daily, oral manner. Imatinib mesylate dose 400 mg/day for pts not on EIAEDs & 1000 mg/day for pts on EIAEDs based on previous studies demonstrating that pts on EIAEDs require significantly higher doses of imatinib mesylate & that such doses are safe & well tolerated. Dose of hydroxyurea 500 mg twice day. Dose level of Zactima will be increased in successive cohorts of pts as described below.
  Cohorts of 3-6 pts will accrue at each dose level until MTD is defined. Each cohort will consist of a mini of 3 newly enrolled pts. Intra-patient dose escalation is not permitted. Cohorts may be expanded at any dose level for further elaboration of safety & pharmacokinetic parameters as required.
  Treatment cycle is defined as daily administration of Zactima + imatinib mesylate & hydroxyurea for 28 days for purpose of scheduling evaluations.
  Other Names: Zactima-ZD6474-Vandetanib; Gleevec-Imatinib mesylate; Hydroxyurea-Droxia-Hydrea-Hydroxycarbamide

SUMMARY:
Primary Objective To determine maximum tolerated dose & dose limiting toxicity of Zactima when combined w standard dosing of imatinib mesylate & hydroxyurea among pts w recurrent malignant glioma who are on & not on enzyme-inducing anti-epileptic drugs Secondary Objectives To assess safety & tolerability of Zactima + imatinib mesylate & hydroxyurea To evaluate pharmacokinetics of Zactima among MG pts on & not on enzyme inducing anti-epileptic drugs (EIAEDs) when combo w imatinib mesylate & hydroxyurea To evaluate pharmacokinetics of imatinib mesylate among MG pts on & not on EIAEDs when combo w Zactima & hydroxyurea Exploratory Objective To evaluate for evidence of anti-tumor activity of study regimen among recurrent malignant glioma (RMG) pts including radiographic response rate, 6-month progression free survival (PFS) rate & median PFS

DETAILED DESCRIPTION:
vascular endothelial growth factor (VEGF) angiogenic & Phosphoinositide 3-kinase inhibitor/Protein Kinase B (PI3K/AKT) mitogenic cascades are 2 upregulated cell signalling pathways in MG that contribute to several hallmark phenotypic features of these tumors. Regimen of Zactima + imatinib mesylate represents novel anti-glioma strategy because it targets 3 key mediators of dysregulated cell signalling involving VEGF & PI3K-AKT pathways including VEGFR, epidermal growth factor receptor (EGFR) & platelet derived growth factor(PDGFR). Furthermore by combining Zactima w imatinib mesylate, VEGF & PI3-k/AKT pathways can potentially inhibit multiple mediators of each of these pathways. Regarding PI3-K/AKT signalling, regimen can inhibit activation of EGFR & PDGFR. Regarding VEGF signalling, regimen has potential to inhibit 3 components of VEGFR directed angiogenesis. 1st, Zactima can directly inhibit VEGFR activation. 2nd, both Zactima & imatinib mesylate can indirectly decrease activity of VEGF pathway by diminishing positive input from activated PI3-K/AKT signalling. 3rd, imatinib mesylate may inhibit PDGF-regulated pericyte maturation of tumor blood vessels.

We have previously demonstrated that regimen of imatinib mesylate + hydroxyurea is active regimen among recurrent glioblastoma multiforme (GBM) pts. Furthermore this activity appears substantially better than that reported for imatinib mesylate alone. Although mechanism of enhanced activity for imatinib mesylate when combo w hydroxyurea is unclear, it is logical to build upon combo of imatinib mesylate + hydroxyurea in subsequent studies rather than imatinib mesylate alone. Current study will therefore determine MTD of Zactima when combo w standard doses of imatinib mesylate & hydroxyurea among RMG pts. Ph II study will then be performed, incorporating maximum tolerated dose (MTD) of Zactima + imatinib mesylate in order to evaluate anti-glioma potential of regimen.

ELIGIBILITY:
Inclusion Criteria:

* Pts have baseline evaluations performed ≤14days prior to 1st dose of study drug unless otherwise specified. Written informed consent must be obtained from pt prior to enrollment
* Pts w MG who are presenting in 1st, 2nd or 3rd recurrence or relapse
* Pts may not have tumor biopsy <1 wk or surgical resection <2wks
* For stratum of non-EIAED pts, each pt be off all EIAEDs for >2 wks prior to starting study drug; similarly for stratum of EIAED pts, each pt be on EIAED for >2 wks prior to starting study drug
* Pts should be on non-increasing dose of steroids for >7 days prior to obtaining baseline Gd-MRI of brain
* Pts should be on non-increasing dose of steroids for >7 days prior to starting study drug
* Multifocal disease is eligible
* Age >18yrs
* Karnofsky Performance Status (KPS) of >70
* Absolute neutrophil count (ANC) > 1.0 x 10 9/L
* Hgb>g/dL
* Platelets>100 x 10 9/L
* Serum creatinine<1.5 x upper limit of normal (ULN)/measured 24hr creatinine clearance (CrCl) >50 milliliters/min/1.73m
* Life ≥12wks
* Written informed consent obtained prior to any screening procedures

Exclusion Criteria:

* Serum bilirubin >1.5x ULN of reference range
* Serum creatinine >1.5 x Upper Limit of the Reference Range (ULRR)/CrCl <50 milliliters/min
* K<4.0 mmol/L despite supplementation; serum Ca/Mg out of normal range despite supplementation
* alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 x ULRR
* Evidence of severe/uncontrolled systemic disease or any concurrent condition which in Investigator's opinion makes it undesirable for pt to participate in trial or which would jeopardize compliance w protocol
* Clinically significant cardiac event such as myocardial infarction; New York Heart Association (NYHA) classification of heart disease >2 within 3 months before entry;/presence of cardiac disease that, in opinion of Investigator, increases risk of ventricular arrhythmia or dysfunction; ejection fraction<50 percent prior to study initiation
* History of arrhythmia-symptomatic/requires treatment/asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is not excluded
* Previous history of corrected QT interval (QTc) prolongation as result from other medication that required discontinuation of that medication
* Congenital long QT syndrome/1st degree relative with unexplained sudden death under 40 years
* Presence of left bundle branch block
* QTc with Bazett's correction that is unmeasurable/>480 msec on screening ECG. If pt has QTc >480 msec on screening ECG, screen ECG may be repeated twice. Average QTc from 3 screening ECGs must be <480 msec in order for pt to be eligible for study
* Any concomitant medication that may cause QTc prolongation, induce Torsades de Pointes/induce cytochrome P450 3A4 (CYP3A4) function except for EIAEDs
* Hypertension not controlled by medical therapy
* Currently active diarrhea that may affect ability of pt to absorb study regimen/tolerate diarrhea
* Pregnant/breast feeding
* Previous/current malignancies of other histologies <1yr, w exception of cervical carcinoma in situ & adequately treated basal cell/squamous cell carcinoma of skin
* Receipt of any investigational agents within 30 days prior to commencing study treatment unless pt has recovered from all anticipated toxicities of investigational agent
* Last dose of prior chemo discontinued <4 wks before start of study therapy unless pt has recovered from all anticipated toxicities of chemo
* Last radiation therapy (XRT) <4wks before start of study therapy, unless pt has recovered from all anticipated toxicities of XRT
* Any unresolved toxicity > Common Terminology Criteria (CTC) grade 1 from previous anti-cancer therapy
* Previous enrollment/randomization of treatment in present study
* Major surgery <4 wks/incompletely healed surgical incision before starting study therapy
* Pts who have received prior oral VEGFR, EGFR/PDGFR-directed therapies
* Pts who are taking warfarin sodium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To determine MTD & dose-limiting toxicity (DLT) & Zactima when combo w Imatinib mesylate & Hydroxyurea among pt w Recurrent MG | 6 months

SECONDARY OUTCOMES:
To further assess safety & tolerability of Zactima & Imatinib mesylate & Hydroxyurea | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, FRCPC, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/